CLINICAL TRIAL: NCT01072240
Title: An Observational Registration Study of Infusion-related Adverse Events at Administration of Mabthera (Rituximab) in the Treatment of Chronic Lymphocytic Leukemia.
Brief Title: An Observational Study on Infusion-related Adverse Events at Administration of MabThera (Rituximab) in Patients With Chronic Lymphocytic Leukemia
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22754
Record Dates: First submitted 2010-02-08; First posted 2010-02-22 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Lymphocytic Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort
  Interventions: Drug: rituximab [Mabthera/Rituxan]

INTERVENTIONS:
Drug: rituximab [Mabthera/Rituxan] — As prescribed by physician

SUMMARY:
This observational study will monitor and register infusion-related adverse events and their handling in patients with chronic lymphocytic leukemia on treatment with MabThera (rituximab). Data will be collected from patients receiving intravenous MabThera at a dose of 375mg/m2 in cycle 1 and 500mg/m2 in subsequent cycles at each treatment visit for up to 6 months. Target sample size is 100 patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >/= 18 years of age
* chronic lymphocytic leukemia treated with rituximab (MabThera)
* rituximab (MabThera) dosage 375 mg/m2 in cycle 1, 500 mg/m2 in subsequent cycles
* informed consent to data collection

Exclusion Criteria:

* participation in an interventional clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CLL patients receiving standard of care rituximab infusions at haematological or medical clinics
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
infusion-related adverse events | data collection every 4-6 weeks for up to 6 months for each patient

SECONDARY OUTCOMES:
usage and applicability of 90-minute iv infusion in patients with CLL | data collection every 4-6 weeks for up to 6 months for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- Sweden (18):
  - Gävle
  - Gothenburg
  - Huddinge
  - Jönköping
  - Kalmar
  - Karlstad
  - Kristianstad
  - Lidköping
  - Linköping
  - Luleå
  - Mora
  - Norrköping
  - Oskarshamn
  - Stockholm
  - Sundsvall
  - Umeå
  - Västervik
  - Visby